CLINICAL TRIAL: NCT02019264
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effect of Long-term Treatment With BELVIQ (Lorcaserin HCl) on the Incidence of Major Adverse Cardiovascular Events and Conversion to Type 2 Diabetes Mellitus in Obese and Overweight Subjects With Cardiovascular Disease or Multiple Cardiovascular Risk Factors
Brief Title: A Study to Evaluate the Effect of Long-term Treatment With BELVIQ (Lorcaserin HCl) on the Incidence of Major Adverse Cardiovascular Events and Conversion to Type 2 Diabetes Mellitus in Obese and Overweight Subjects With Cardiovascular Disease or Multiple Cardiovascular Risk Factors
Acronym: CAMELLIA-TIMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD356-G000-401; 2013-000324-34 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Disease; High Cardiovascular Risk; Obesity; Overweight; Type 2 Diabetes
Keywords: Diabetes; Cardiovascular Disease; Multiple Cardiovascular Risk Factors; Obesity; Overweight; MACE; Conversion to Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Overweight; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Lorcaserin hydrochloride (HCL)10 mg (Experimental): APD356 10 mg twice daily
  Interventions: Drug: Lorcaserin hydrochloride
- Placebo (Placebo Comparator): Placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin hydrochloride — APD356 10 mg twice daily
  Other Names: APD356; BELVIQ
  Arms: Lorcaserin hydrochloride (HCL)10 mg
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study in overweight and obese subjects with cardiovascular (CV) disease and/or multiple CV risk factors.

DETAILED DESCRIPTION:
Approximately 12,000 subjects will be randomized to two treatment groups in a ratio of 1:1, stratified by the presence of established CV disease (approximately 80%) or CV risk factors without established CV disease (approximately 20%). Subjects will receive lorcaserin HCl 10 mg BID or placebo BID. The study will consist of 2 phases: Prerandomization and Randomization. The Prerandomization Phase will last up to 30 days and consist of one visit during which subjects will be screened for eligibility. The Randomization Phase will consist of two periods: Treatment and Follow-up. The Treatment Period will last for approximately 5 years with approximately 18 visits and Follow-up period is 30 (+ or - 10 days) from the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria

1. BMI greater than or equal (>=) to 27 kilogram per meter square (kg/m^2)
2. Subjects able and willing to comply with a reduced-calorie diet and an increased physical activity program
3. Age >= to 40 years with established CV disease as defined by one of the following:

   1. History of documented MI or ischemic stroke
   2. History of peripheral artery disease
   3. History of revascularization (coronary, carotid, or peripheral artery)
   4. Significant unrevascularized coronary arterial stenosis

OR

Age >= to 55 years for women or >= to 50 years for men who have type 2 diabetes mellitus (T2DM) without established CV disease plus at least one of the following CV risk factors:

1. Hypertension, or currently receiving therapy for documented hypertension
2. Dyslipidemia, or currently taking prescription lipid-lowering therapy for documented dyslipidemia
3. Estimated glomerular filtration rate >= to 30 to less than equal (<=) to 60 mililitre per minute per 1.73 meter square (mL/min/1.73 m^) per the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
4. High high sensitivity C-reactive protein (hsCRP)
5. Urinary albumin-to-creatinine ratio (ACR) >= 30 ug/mg

Subjects with T2DM may have a pre-existing or new diagnosis of T2DM. A new diagnosis of T2DM (ie, discovered at Screening) should be based on the 2013 American Diabetes Association (ADA) guidelines.

All T2DM subjects must have an HbA[1c] less (<) than 10% at Screening. If subjects are being treated, or upon diagnosis need to be treated with antidiabetic agents, the T2DM treatment regimen must be stable for at least 3 months prior to randomization.

Exclusion Criteria

1. Moderate or greater symptoms of congestive cardiac failure (New York Heart Association [NYHA] class III or IV)
2. Known left ventricular (LV) ejection fraction < than 20%
3. Moderate or greater symptoms of pulmonary hypertension (PH)
4. Known severe valvular disease
5. Moderate renal impairment, severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m^ per the CKD-EPI equation based on ideal body weight), or end stage renal disease (ESRD)
6. Severe hepatic impairment
7. Use of other products intended for weight loss including prescription drugs, over-the-counter (OTC) drugs, and herbal preparations
8. Use of more than one other serotonergic drug
9. Use of drugs known to increase the risk for cardiac valvulopathy within 6 months prior to Screening including, but not limited to: pergolide, ergotamine, methysergide, cabergoline
10. History or evidence of clinically significant disease (e.g., malignancy, cardiac, respiratory, gastrointestinal, renal or psychiatric disease)
11. Use of lorcaserin HCl prior to Screening or hypersensitivity to lorcaserin HCl or any of the excipients
12. Planned bariatric surgery
13. Females must not be breastfeeding or pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14673 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (498):
- United States (372):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - UAB Medical Center, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Connect Clinical Research Center, LCC, Chandler, Arizona
  - Arrowhead Health Centers, Glendale, Arizona
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Arkansas Cardiology Clinic, Little Rock, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Preferred Research Partners, Little Rock, Arkansas
  - Clinical Research Alliance, Alhambra, California
  - Central Cardiology, Bakersfield, California
  - Cardiovascular Research Foundation of Southern Cal, Beverly Hills, California
  - Capitol Interventional Cardiology, Carmichael, California
  - San Diego Costal Endocrinology Group AMC, Chula Vista, California
  - John Muir Physician Network Clinical Research Cent, Concord, California
  - Medical Group of Encino, Encino, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - California Heart Specialists, Huntington Beach, California
  - Del Rosario Medical Clinic, Inc., Huntington Park, California
  - Diabetes and Endocrine Associates, La Mesa, California
  - La Mesa Cardiac Center, La Mesa, California
  - Alliance Research Centers, Laguna Hills, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Metabolic Clinic and Research Center, Los Angeles, California
  - Beverly Hills Cardiology, Los Angeles, California
  - VA Greater Los Angeles Health Care System, Los Angeles, California
  - Clinical Interventions Research Institute, Mission Viejo, California
  - Brigid Freyne MD Inc, Murrieta, California
  - Valley Clinical Trials Inc, Northridge, California
  - Carr Cardiology, Oceanside, California
  - Northern California Clinical Research Center, Redding, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - University of California San Diego, San Diego, California
  - Ritchken and First MD's, San Diego, California
  - West Coast Research LLC, San Ramon, California
  - Coastal Multi-Specialty Research, Santa Ana, California
  - Westlake Medical Research, Thousand Oaks, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Ronald Chochinov, MD, Ventura, California
  - Ventura Cardiology Consultants, Ventura, California
  - Infosphere Clinical Research, West Hills, California
  - UCH-MHS Cardiac Research, Colorado Springs, Colorado
  - Creekside Endocrine Associates PC, Denver, Colorado
  - New West Physicians, PC, Golden, Colorado
  - University of Colorado Health, Loveland, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Clinical Research Works, Bristol, Bristol, Connecticut
  - Cardiology Associates of Fairfield County, Norwalk, Norwalk, Connecticut
  - Cardiology Associates of Fairfield County, P.C., Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Cardiology Associates of Fairfield County, P.C., Trumbull, Connecticut
  - Connecticut Heart and Vascular Center, Trumbull, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Red Clay Research, Newark, Delaware
  - Alfieri Cardiology, Wilmington, Delaware
  - Aventura Heart Center, Aventura, Florida
  - Zasa Clinical Research, Boynton Beach, Florida
  - Meridien Research, Bradenton, Florida
  - NOVA Southeastern University, Bradenton, Florida
  - Bay Area Cardiology, Brandon, Florida
  - Meridien Research, Brooksville, Brooksville, Florida
  - Clearwater Cardiovascular and Interventional Cons., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Holy Cross Medical Group, Coral Springs, Florida
  - Cardiology Research Associates, Daytona Beach, Florida
  - International Medical Research, Daytona Beach, Florida
  - Asclepius Medical Research, Doral, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Integrative Research Associates, Inc., Fort Lauderdale, Florida
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Primary Care Associates, Fort Myers, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - George E. Platt, M.D., Green Cove Springs, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - Larry K. Levinson, D.O., P.A., Hollywood, Florida
  - Research Physicians Network Alliance, Hollywood, Florida
  - Pasco Cardiology Center, Hudson, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - University of Florida- Jacksonville, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Pharmax Research Clinic, Inc, Miami, Florida
  - Life Spring Research Foundation, Miami, Florida
  - United Clinical Research Corp., Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - South Florida Research Group LLC, Miami, Florida
  - South Florida Research Solutions, Miramar, Florida
  - Southwest Florida Research, Naples, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Palm Beach Gardens Research Center, Palm Beach Gardens, Florida
  - Research Physicians Network Alliance, Pembrok, Pembroke Pines, Florida
  - South Florida Research Solutions, Pembroke Pines, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Columbia Primary Care, LLC d/b/a Heart and Health Institute, Plantation, Florida
  - St Johns Center for Clinical Research, Ponte Vedra, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Brevard Cardiovascular Research Associates Inc, Rockledge, Florida
  - Clearwater Cardiovascular and Interventional Cons., Safety Harbor, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Springfield Medical Center, Springfield, Florida
  - Bayfront Health St. Petersburg, Research, St. Petersburg, Florida
  - Meridien Research - St. Petersburg, St. Petersburg, Florida
  - Professional Health Care of Pinellas, INC, St. Petersburg, Florida
  - Advanced Clinical Research Group, Stuart, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Healthpoint Medical Group, Inc, Tampa, Florida
  - Interventional Cardiac Consultants, Trinity, Florida
  - Lovelace Scientific Research, Venice, Florida
  - Indian River Medical Center-Cardiology, Vero Beach, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cleveland Clinic Foundation, West Palm Beach, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Diabetes Associates, Endocrinology, Atlanta, Georgia
  - Rockdale Medical-Research Associates, Conyers, Georgia
  - Atlanta Heart Specialists, Cumming, Georgia
  - Urban Family Practice Associates/Clinical Research Advantage, Marietta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Herman Clinical Research LLC, Suwanee, Georgia
  - Atlanta Heart Specialists, Tucker, Georgia
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Consultants in Cardiovascular Medicine, Elmhurst, Illinois
  - Clinical Investigation Specialists, Inc. in Gurnee, Gurnee, Illinois
  - Advanced CardioVascular Consultants, SC, Rock Island, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - American Health Network of IN, LLC, Avon, Avon, Indiana
  - Premier Healthcare, LLC, Bloomington, Indiana
  - Deaconess Clinic, Inc., Evansville, Indiana
  - American Health Network of IN, LLC, Franklin, Franklin, Indiana
  - American Health Network of IN, LLC, Greenfield, Greenfield, Indiana
  - American Health Network - Thomas Moretto, MD, Indianapolis, Indiana
  - Medical Consultants PC, Muncie, Indiana
  - American Health Network of IN, LLC, Muncie, Indiana
  - Cardiology Associates of Northwest Indiana, P.C, Munster, Indiana
  - The University of Iowa, College of Public Health, Iowa City, Iowa
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Norton Heart Specialists, Louisville, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Research Integrity LLC, Owensboro, Kentucky
  - Central Maine Medical Center, Auburn, Maine
  - Acadia Clinical Research, LLC, Bangor, Maine
  - Eastern Maine Medical Center Northeast Cardiology Associates, Bangor, Maine
  - Southern Maine Health Care/Maine Medical Center Research Ins, Biddeford, Maine
  - InterMed, PA, Portland, Maine
  - Medstar Cardiology Associates, Annapolis, Maryland
  - Chesapeake Cardiovascular Associates, GBMC, Baltimore, Maryland
  - Clinical Research, Inc, Baltimore, Maryland
  - Medstar Union Memorial Heart Specialists, Baltimore, Maryland
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Spectrum Clinical Research, Baltimore, Maryland
  - Overlea Personal Physicians, Baltimore, Maryland
  - Shahid Saeed MD, PC, Baltimore, Maryland
  - Maryland Heart Associates, LLC, Glen Burnie, Maryland
  - Klein & Associates, MD, PA, Hagerstown, Maryland
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Lutherville Personal Physicians, Lutherville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Endocrine & Metabolic Consultants, Rockville, Maryland
  - Lutherville Personal Physicians, Towson, Maryland
  - Overlea Personal Physicians, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - MGH Weight Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New England Center for Clinical Research, IMCA, Fall River, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - ActivMed Practices, Methuen, Massachusetts
  - Partners Community Physicians Organization, Natick, Massachusetts
  - Partners Community Physicians Organization, Needham, Massachusetts
  - Endeavor Medical Research PLC, Alpena, Michigan
  - Cadillac Clinical Research, LLC, Cadillac, Michigan
  - Westside Family Medical Center, PC, Kalamazoo, Michigan
  - Cardiology Consultants of East Michigan, Lapeer, Michigan
  - Marquette General Heart and Vascular Institute, Marquette, Michigan
  - MidMichigan Medical Center, Midland, Michigan
  - Nisus Research at McLaren Northern Michigan Hospital, Petoskey, Michigan
  - Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Remedica LLC, Rochester, Michigan
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - American Center for Clinical Trials, Southfield, Michigan
  - Medical Research Associates, Inc., Traverse City, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Baxter, Minnesota
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - MNCOME Clinic, Eagan, Minnesota
  - Radiant Research, Inc., Edina, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Coast Cardiovascular Consultants PLLC, Gulfport, Mississippi
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Diabetes & Endocrinology Specialists, Inc., Chesterfield, Missouri
  - BodyAesthetic Research Center, Washington, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Montana Health Research Institute, Inc., Billings, Montana
  - Glacier View Cardiology PC, Kalispell, Montana
  - Internal Medical Associates of Grand Island, PC, Grand Island, Nebraska
  - Clinical Research Advantage / Rita Chuang, M.D., Henderson, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Medicor Cardiology, PA, Bridgewater, New Jersey
  - Advanced Heart Care, Bridgewater, New Jersey
  - UmiMed Center LLC, East Brunswick, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Elmer, New Jersey
  - Advocare Heights Primary Care, Haddon Heights, New Jersey
  - Cardiovascular Associates of the Delaware Valley P, Haddon Heights, New Jersey
  - NJ Heart, Linden, New Jersey
  - Rutgers New Jersey Medical School, Mine Hill, New Jersey
  - Cardiovascular Associates Delaware Valley Sewell, Sewell, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Albany College of Medicine, Division of Endocrinology, Albany, New York
  - Capital Cardiology Associates, Albany, New York
  - United Medical Associates, PC, Binghamton, New York
  - Buffalo Heart Group, Buffalo, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Long Island Heart Associates, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - DiGiovanna Institute for Medical Education, North Massapequa, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Northwell Health Physician Partners Cardiology, Southampton, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Capital Cardiology Associates, Troy, New York
  - Great Lakes Medical Research, Westfield, New York
  - Kernodle Clinic, Burlington, North Carolina
  - Clinical Trials of America Inc., Cary, North Carolina
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Bland Clinic, PA, Greensboro, North Carolina
  - Clinical Trials of America Inc. Hickory, Hickory, North Carolina
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Clinical Trials of America, Inc., Lenoir, North Carolina
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Rocky Mount, Rocky Mount, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Aultman Hospital, Canton, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Sentral Clinical Research, Cincinnati, Ohio
  - Delaware Research Group, LLC, Delaware, Ohio
  - Awasty Research Network, LLC, Marion, Ohio
  - Community Health Care, Massillon, Ohio
  - Apex Medical Research Inc., Springfield, Ohio
  - Integris Cardiovascular Physicians LLC, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute PC, Tulsa, Oklahoma
  - Blair Medical Associates, Altoona, Pennsylvania
  - Clinical Research Associates of Central PA, LLC, Altoona, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Geisinger Health Clinic, Danville, Pennsylvania
  - Geisinger Health System, Danville, Pennsylvania
  - Doylestown Health Cardiology a Division of Doylestown Health, Doylestown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Liberty Family Practice, Erie, Pennsylvania
  - Endocrine Clinical Research LLC, Feasterville, Pennsylvania
  - Joseph Lamantia, DO, Indiana, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Lycoming Internal Medicine, Inc., Jersey Shore, Pennsylvania
  - Berkley Hills Clinicals, Johnstown, Pennsylvania
  - Ilumina Clinical Associates, Johnstown, Johnstown, Pennsylvania
  - Joseph Lamantia, DO, Johnstown, Pennsylvania
  - Comprehensive Cardiology Consultants, Langhorne, Pennsylvania
  - Detweiler Family Medicine and Associates PC, Lansdale, Pennsylvania
  - Green & Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Capital Area Research LLC, Newport, Pennsylvania
  - Endocrine Metabolic Associates, Philadelphia, Pennsylvania
  - Pottstown Medical Specialists, Inc. (PMSI), Pottstown, Pennsylvania
  - Geisinger Clinic, Scranton, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Radiant Research, Inc., Greer, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Palmetto Research Center, LLC, Spartanburg, South Carolina
  - Brown Clinic, PLLP, Watertown, South Dakota
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Chattanooga Research and Medicine (CHARM), Chattanooga, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Wellmont CVA Heart Institute, Greeneville, Tennessee
  - Research Associates of Jackson, Jackson, Tennessee
  - Kore Cardiovascular Research, Jackson, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Wellmont CVA Heart Institute, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - The Endocrine Clinic, Memphis, Tennessee
  - Cardiology Wellness Center, Nashville, Tennessee
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Texas Health Physicians Group, Carrollton, Texas
  - Adriana Pop-Moody MD Clinic, PA, Corpus Christi, Texas
  - Baylor Research Institute, Dallas, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - Texas Health Physicians Group, Dallas, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Odilon Alvarado, M.D., Fort Worth, Texas
  - Texas Health Physicians Group Fort Worth, Fort Worth, Texas
  - Tand R Clinic, PA, Fort Worth, Texas
  - San Gabriel Clinical Research, LLC, Georgetown, Texas
  - Angiocardiac Care of Texas PA, Houston, Texas
  - Oxford Clinical Research, LLC, Houston, Texas
  - West Houston Area Clinical Trial Consultants, LLC, Houston, Texas
  - Endocrine and Psychiatry Center, Houston, Texas
  - Texas Health Physicians Group, Irving, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Jalil Aziz Khan M.D., P.A., Lewisville, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Permian Research Foundation, Odessa, Texas
  - Medical Clinic of North Texas, Plano, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Texas Diabetes, Round Rock, Texas
  - Physician PrimeCare Research Institute, PLLC, San Antonio, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Bay Area Total Health Medical Group, Webster, Texas
  - Advanced Research Institute, Ogden, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Alexandria Clinical Research, LLC, Alexandria, Virginia
  - Washington Center for Weight Management and Resear, Arlington, Virginia
  - Burke Internal Medicine and Research, Burke, Virginia
  - Cardiology Consultants of Danville, Inc., Danville, Virginia
  - Danville Internal Medicine, Inc, Danville, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Seven Corners Medical Research Center, Falls Church, Virginia
  - INOVA Health Care Services, Manassas, Virginia
  - Burke Internal Medicine and Research, Manassas, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Health Research of Hampton Roads - Norfolk, Inc., Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Clinical Research Partners, Richmond, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - National Clinical Research-Richmond, Inc, Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Larry D. Stonesifer, MD, Inc PS, Federal Way, Washington
  - Seattle Women's, Seattle, Washington
  - Rowan Research Inc., Spokane, Washington
  - MultiCare Research Institute, Tacoma, Washington
  - Universal Research Group, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Cardiology Associates of Bellin Health, Green Bay, Wisconsin
  - Prevea Clinic, Inc, Green Bay, Wisconsin
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
  - Meriter hospital Inc., DBA: UnityPoint Health-Meriter Heart, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aspirus Research Institute, Wausau, Wisconsin
- Australia (23):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Gosford Hospital, Cardiology Clinical Trials, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Illawarra Shoalhaven Local Health District, Clinical Trial and Research Unit, Wollongong, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Core Research Group, Brisbane, Queensland
  - Princess Alexandra Hospital, Cardiology Research Department, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Endocrinology Department, Herston, Queensland
  - HeartCare Partners Clinical Research Unit, Milton, Queensland
  - AusTrials Pty Ltd, Sherwood, Queensland
  - Gold Coast Hospital, Cardiovascular Research Centre, Southport, Queensland
  - New Royal Adelaide Hospital, Cardiology Department, Adelaide, South Australia
  - Adelaide Medical Research, Ashford, South Australia
  - Lyell McEwin Hospital, Department of Cardiology, Elizabeth Vale, South Australia
  - Heart and Vascular Institute, Fullarton, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Health Services, Ballarat, Victoria
  - Geelong Cardiology Research Unit, Barwon Health, Geelong, Victoria
  - Austin Health - Heidelberg Repatriation Hospital, Department of Medicine, Boronia Centre, Heidelberg Heights, Victoria
  - Avenue Cardiovascular Centre, Saint Kilda East, Victoria
  - Joondalup Cardiovascular Trials Foundation Inc, Joondalup, Western Australia
  - Fiona Stanley Hospital, Cardiology Research Department,CDO11, Murdoch, Western Australia
  - South Australian Medical Research Inst, Centre for Clinical Research, Adelaide
- Canada (38):
  - LMC Clinical Research Inc. (Calgary), Calgary, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Nova Scotia Health Authority /QEII Health Sciences Centre, Halifax, Nova Scotia
  - LMC Diabetes & Endocrinology - Brampton, Brampton, Ontario
  - McMaster University, Brampton, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - Aviva Clinical Trial Group In., Burlington, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Joanne F. Liutkus Medicine Professional Corp., Cambridge, Ontario
  - Saul Vizel Professional Medicine Corporation, Vizel Cardiac Research, Cambridge, Ontario
  - LMC Diabetes & Endocrinology (Etobicoke), Etobicoke, Ontario
  - Dr. Dinkar Shukla Professional Medicine Corporation, Greater Sudbury, Ontario
  - Dr Roger Labonte Professional Medicine Corp, Greater Sudbury, Ontario
  - Wharton Medical Clinic Clinical Trials Group Inc., Hamilton, Ontario
  - Saint Josephs Health Care London, London, Ontario
  - LMC Diabetes & Endocrinoly, Markham, Ontario
  - New Market Cardiology Research Group, Newmarket, Ontario
  - Dr. Michael Heffernan, Oakville, Ontario
  - LMC Clinical Research Inc. (Oakville), Oakville, Ontario
  - Dr. Cha, Oshawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - LMC Diabetes & Endocrinology (Thornhill), Thornhill, Ontario
  - JJ DIG Research Ltd., Toronto, Ontario
  - Keele Medical Place, Toronto, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - St Michael's Hospital Health Centre, Toronto, Ontario
  - ViaCar Recherche Clinique, Brossard, Quebec
  - Q&T Research Outaouais Inc., Gatineau, Quebec
  - ViaCar Recherche Clinique Inc., Greenfield Park, Quebec
  - Manna Research Inc, Lévis, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
  - Centre hospitalier régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - CardioVasc HR, Inc., Saint-Jean-sur-Richelieu, Quebec
  - ViaCar Recherche Clinique Inc., Saint-Lambert, Quebec
  - LMC Clinical Research Inc. (Montreal), Saint-Laurent, Quebec
  - Recherche Clinique London, Sherbrooke, Quebec
- Chile (8):
  - Biomedica Research Group, Providencia, Santiago Metropolitan
  - Sociedad Medica Cardiologica El Llano, San Miguel, Santiago Metropolitan
  - Hospital Regional Concepcion, Concepción
  - Cardiocob, Santiago
  - Servicios Medicos Godoy Ltda., Santiago
  - Ccbr Cecim, Santiago
  - Centro Investigacion Clinica del Sur, Temuco
  - CECMI Ltda., Temuco
- Mexico (9):
  - ICLE, Guadalajara, Jalisco
  - Private Medical Practice, Guadalajara, Jalisco
  - IMED Clin Trials, Monterrey, Nuevo León
  - Cardiolink ClinTrials S.C., Monterrey, Nuevo León
  - Centro de Estudios Clinicos y Especialidades Medicas S.C., Monterrey, Nuevo León
  - Hospital de Angeles Xalapa, Xalapa, Veracruz
  - Fundacion Cardiovascular de Aguascalientes, Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Mentrials S.A.de C.V., Distrito Federal
- New Zealand (13):
  - North Shore Hospital-Cardiology Research, Milford, Auckland
  - Middlemore Hospital, Papatoetoe, Auckland
  - North Shore Hospital - Diabetes Clinic, Takapuna, Auckland
  - Christchurch Hospital, Lipids, Christchurch, Canterbury
  - Christchurch Hospital, Cardiology Research, Christchurch, Canterbury
  - Dunedin Hospital, Dunedin, Otago
  - Taranaki Base Hospital, New Plymouth, Taranaki Region
  - Hutt Hospital, Cardiology Dept, Lower Hutt, Wellington Region
  - Auckland City Hospital, Auckland
  - Hawkes Bay Regional Hospital, Hastings
  - Nelson Hospital, Cardiology Department, Nelson
  - Lakeland Clinical Trials, Rotorua, Rotorua
  - Tauranga Hospital, Tauranga
- Poland (34):
  - Indywidualna Specjalistyczna Praktyka Lekarska, Bezrzecze
  - Podlaski Osrodek Kardiologii Janusz Korecki, Bialystok
  - NZOZ "Eskulap", Biała Rawska
  - Centrum Medyczne KERmed, Bydgoszcz
  - 10 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ, Bydgoszcz
  - Nzoz "Mada-Med", Chorzów
  - DIABET Centrum Medyczne s. c., Chrzanów
  - ISPL w Dziedzinie Kardiologii lek.med. Krzysztof Cymerman, Gdynia
  - NZOZ SCBK ProCordis, Gdynia
  - Gabinet Kardiologiczno-Internistyczny, Gdynia
  - Praktyka Lekarska dr n. med. Marek Bronisz, Inowrocław
  - Piotr Mader Diabetic Clinic NZOZ PD-I, Kamieniec Ząbkowicki
  - NZOZ Eskulap SC, Koluszki
  - Ewa Mirek-Bryniarska Specjalistyczna Praktyka Lekarska, Krakow
  - LANDA' Specjalistyczne Gabinety Lekarskie, Krakow
  - Medyczne Centrum Diabetologiczno Endokrynologiczno, Krakow
  - Nzoz Cardiamed, Legnica
  - NZOZ ALL-MED Centrum Medyczne, Lodz
  - "CenterMed Lublin" Sp. z o.o., Lublin
  - Indywidualna Praktyka Lekarska, Mrągowo
  - Zechowicz MEDEUSZ-PLUS, Olsztyn
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - NZOZ NEURO-KARD "Ilkowski i Partnerzy", Poznan
  - Specjalistyczna Przychodnia Lekarska MEDIKARD (SPL Medikard), Płock
  - Specjalistyczny Gabinet Lekarski, Tarnów
  - Lecznice Citomed Sp. z o.o., Torun
  - Praktyka Lekarska Pawlowicz Lidia, Torun
  - Centrum Medyczne AMED, Warsaw
  - Centrum Badawcze Wspolczesnej Terapii, Warsaw
  - SNZOZ Fundacji PROCLINICA, Warsaw
  - Centrum Zdrowia Wierzchoslawice, Wierzchosławice
  - Regionalna Poradnia Diabetologiczna, Wroclaw
  - Specjalistyczne Gabinety Lekarskie "Medicor PLUS", Włocławek
  - SP ZOZ w Lecznej, Łęczna
- The Partners Clinical Research Centre, Nassau, The Bahamas

REFERENCES:
- [Derived] Scirica BM, Bohula EA, Dwyer JP, Qamar A, Inzucchi SE, McGuire DK, Keech AC, Smith SR, Murphy SA, Im K, Leiter LA, Gupta M, Patel T, Miao W, Perdomo C, Bonaca MP, Ruff CT, Sabatine MS, Wiviott SD; CAMELLIA-TIMI 61 Steering Committee and Investigators. Lorcaserin and Renal Outcomes in Obese and Overweight Patients in the CAMELLIA-TIMI 61 Trial. Circulation. 2019 Jan 15;139(3):366-375. doi: 10.1161/CIRCULATIONAHA.118.038341. PMID 30586726
- [Derived] Bohula EA, Scirica BM, Inzucchi SE, McGuire DK, Keech AC, Smith SR, Kanevsky E, Murphy SA, Leiter LA, Dwyer JP, Corbalan R, Hamm C, Kaplan L, Nicolau JC, Ophuis TO, Ray KK, Ruda M, Spinar J, Patel T, Miao W, Perdomo C, Francis B, Dhadda S, Bonaca MP, Ruff CT, Sabatine MS, Wiviott SD; CAMELLIA-TIMI 61 Steering Committee Investigators. Effect of lorcaserin on prevention and remission of type 2 diabetes in overweight and obese patients (CAMELLIA-TIMI 61): a randomised, placebo-controlled trial. Lancet. 2018 Nov 24;392(10161):2269-2279. doi: 10.1016/S0140-6736(18)32328-6. Epub 2018 Oct 4. PMID 30293771
- [Derived] Bohula EA, Wiviott SD, McGuire DK, Inzucchi SE, Kuder J, Im K, Fanola CL, Qamar A, Brown C, Budaj A, Garcia-Castillo A, Gupta M, Leiter LA, Weissman NJ, White HD, Patel T, Francis B, Miao W, Perdomo C, Dhadda S, Bonaca MP, Ruff CT, Keech AC, Smith SR, Sabatine MS, Scirica BM; CAMELLIA-TIMI 61 Steering Committee and Investigators. Cardiovascular Safety of Lorcaserin in Overweight or Obese Patients. N Engl J Med. 2018 Sep 20;379(12):1107-1117. doi: 10.1056/NEJMoa1808721. Epub 2018 Aug 26. PMID 30145941
- [Derived] Bohula EA, Scirica BM, Fanola C, Inzucchi SE, Keech A, McGuire DK, Smith SR, Abrahamsen T, Francis BH, Miao W, Perdomo CA, Satlin A, Wiviott SD, Sabatine MS. Design and rationale for the Cardiovascular and Metabolic Effects of Lorcaserin in Overweight and Obese Patients-Thrombolysis in Myocardial Infarction 61 (CAMELLIA-TIMI 61) trial. Am Heart J. 2018 Aug;202:39-48. doi: 10.1016/j.ahj.2018.03.012. Epub 2018 Mar 29. PMID 29803985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites in the United States, Bahamas, Canada, Mexico, Chile, New Zealand, Poland, and Australia from 24 Jan 2014 to 14 May 2018.
Pre-assignment Details: A total of 14,673 participants were screened and enrolled, of which 2673 participants were screen failures and 12,000 were randomized to receive lorcaserin hydrochloride (HCl) or placebo.
Groups:
- Placebo: Participants received lorcaserin HCL placebo-matching, tablets, orally, twice daily for up to 52 months.
- Lorcaserin 10 mg: Participants received lorcaserin HCL 10 milligram (mg), tablets, orally, twice daily for up to 52 months.
Period: Overall Study
Arm/Group | Placebo | Lorcaserin 10 mg
Started | 6000 | 6000
Safety Analysis Set | 5992 | 5995
Completed (Participants who died on trial were considered completed.) | 5752 | 5793
Not Completed | 248 | 207
Not completed — Not treated | 6 | 4
Not completed — Lost to Follow-up | 50 | 47
Not completed — Withdrawal by Subject | 142 | 117
Not completed — Administrative reason | 36 | 28
Not completed — Missing | 14 | 11

BASELINE CHARACTERISTICS:
Population: The full analysis (FA) set included all randomized participants regardless of whether they took study drug or not.
Groups:
- Lorcaserin 10 mg: Participants received lorcaserin HCL 10 mg, tablets, orally, twice daily for up to 52 months.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lorcaserin 10 mg | Total
Number analyzed (Participants) | 6000 | 6000 | 12000
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.31) | 63.5 (8.33) | 63.6 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2186 | 2112 | 4298
  Male | 3814 | 3888 | 7702
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 536 | 502 | 1038
  Not Hispanic or Latino | 5464 | 5498 | 10962
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 26 | 47
  Asian | 74 | 85 | 159
  Native Hawaiian or Other Pacific Islander | 23 | 30 | 53
  Black or African American | 466 | 454 | 920
  White | 5331 | 5309 | 10640
  More than one race | 85 | 96 | 181
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to First Occurrence of Major Adverse Cardiovascular Events (MACE) at Interim Analysis
Description: The MACE events involved myocardial infarction (MI), stroke, or cardiovascular (CV) death. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to Month 42
Population: The total time analysis set using the intent-to-treat (ITT) set, events were counted that occurred while participants were on and off treatment. Participants with no events were censored at their last study contact or at the visit following sponsor notification of study completion, whichever occurred first.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 6000 | 6000
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Non-Inferiority — Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates. MACE met non-inferiority when the one-sided upper bound of 97.5% confidence interval of the HR was less than 1.4 (the non-inferiority margin); p = 0.0001, Primary Analytic Method; Hazard Ratio (HR) = 1.005, 97.5% CI 2-sided [0.842 to 1.198]

2. Primary Outcome: Time From Randomization to First Occurrence of MACE+
Description: The MACE+ events involved MI, stroke, or CV death or hospitalization for unstable angina or heart failure (HF), or any coronary revascularization. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The total time analysis set used the ITT set, events were counted that occurred while participants were on and off treatment. Participants with no events were censored at their last study contact or at the visit following Sponsor Notification of Study Completion, whichever occurred first.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 6000 | 6000
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.5464, Primary Analytic Method; Hazard Ratio (HR) = 0.969, 95% CI 2-sided [0.873 to 1.074]

3. Secondary Outcome: Time From Randomization to Conversion to Type 2 Diabetes Mellitus (T2DM) for Participants With Prediabetes at Baseline
Description: Time from randomization to conversion to T2DM was defined as first occurrence of any component of the 2013 American Diabetes Association (ADA) Diagnostic Criteria (ADA, 2013) in participants with prediabetes at baseline. The diagnostic criteria were met if a participant had unequivocal hyperglycemia (random plasma glucose greater than or equal to (>=) 200 milligram per deciliter (mg/dL) (11.1 millimole per liter [mmol/L]) with classic symptoms of hyperglycemia or hyperglycemic crisis) or any of the following criteria were observed and subsequently confirmed on repeat laboratory testing such as: glycosylated hemoglobin (HbA1c) >=to 6.5%; fasting plasma glucose (FPG) >=126 mg/dL (7.0 mmol/L); 2-hour plasma glucose >=200 mg/dL (11.1 mmol/L) by an oral glucose tolerance test (OGTT). The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: Prediabetes and total time analysis set used ITT set: without a history of any type of diabetes and who were prediabetic at baseline; events were counted that occurred while participants were on, off treatment; participants with no events were censored at last study contact/at visit after notification of study completion, whichever occurred first.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 1976 | 2015
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on Cox-regression model including treatment as covariate; p = 0.0380, Primary Analytic Method; Hazard Ratio (HR) = 0.807, 95% CI 2-sided [0.659 to 0.988]

4. Secondary Outcome: Time From Randomization to First Occurrence of the Individual Components of MACE+
Description: The MACE+ events involved MI, stroke, or CV death or hospitalization for unstable angina or HF, or any coronary revascularization. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The total time analysis set used the ITT set, events counted occurred while participants were on and off treatment. Participants with no events were censored at last study contact or at the visit following Sponsor Notification of Study Completion, whichever first.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 6000 | 6000
days
  MI | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
  Stroke | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
  CV death | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
  Hospitalization for unstable angina | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
  HF | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
  Coronary revascularization | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Non-Inferiority — Myocardial Infarction: Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates. 97.5% confidence interval refers to the upper limit of the displayed 2-sided 95% confidence interval; p = 0.0001, Primary Analytic Method; Hazard Ratio (HR) = 0.991, 97.5% CI 2-sided [0.824 to 1.191]
Statistical Analysis 2: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Non-Inferiority — Time to Stroke: Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates. 97.5% CI refers to the upper limit of the displayed 2-sided 95% CI; p = 0.0005, Primary Analytic Method; Hazard Ratio (HR) = 0.856, 97.5% CI 2-sided [0.639 to 1.145]
Statistical Analysis 3: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Non-Inferiority — Cardiovascular Death: Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates. 97.5% confidence interval refers to the upper limit of the displayed 2-sided 95% confidence interval; p = 0.0262, Primary Analytic Method; Hazard Ratio (HR) = 1.045, 97.5% CI 2-sided [0.778 to 1.404]
Statistical Analysis 4: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hospitalization for Unstable Angina: Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.3243, Primary Analytic Method; Hazard Ratio (HR) = 1.163, 95% CI 2-sided [0.861 to 1.571]
Statistical Analysis 5: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Heart Failure: Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.6758, Primary Analytic Method; Hazard Ratio (HR) = 0.952, 95% CI 2-sided [0.757 to 1.197]
Statistical Analysis 6: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Coronary Revascularization: Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.7817, Primary Analytic Method; Hazard Ratio (HR) = 0.981, 95% CI 2-sided [0.856 to 1.125]

5. Secondary Outcome: Time From Randomization to Event of All-cause Mortality
Description: The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 6000 | 6000
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.4212, Primary Analytic Method; Hazard Ratio (HR) = 1.082, 95% CI 2-sided [0.893 to 1.310]

6. Secondary Outcome: Time From Randomization to Conversion to Normal Glucose Homeostasis in Participants With Prediabetes at Baseline
Description: Normal glucose homeostasis was defined as HbA1c less than or equal to (<=) 5.6% and FPG < 100 mg/dL without any antidiabetic treatment. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The prediabetes analysis set included all participants in the ITT set without a history of any type of diabetes and who were prediabetic at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 1976 | 2015
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on a Cox regression model including treatment as covariate; p = 0.1810, Primary Analytic Method; Hazard Ratio (HR) = 1.124, 95% CI 2-sided [0.947 to 1.333]

7. Secondary Outcome: Time From Randomization to Conversion to T2DM for Participants Without Any Type of Diabetes at Baseline
Description: The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The nondiabetes analysis set included all participants in the ITT set without a history of any type of diabetes at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 2569 | 2615
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on a Cox regression model including treatment as covariate; p = 0.0116, Primary Analytic Method; Hazard Ratio (HR) = 0.773, 95% CI 2-sided [0.633 to 0.944]

8. Secondary Outcome: Change From Baseline in HbA1c at Month 6 in Participants With T2DM at Baseline
Time Frame: Baseline, and Month 6
Population: The T2DM analysis set included all participants in the ITT set who had T2DM at baseline. The T2DM analysis set where data was available at specified time points.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 3403 | 3362
percentage of HbA1c
  Baseline | 6.99 (1.066) | 7.01 (1.082)
  Change at Month 6: number analyzed (Participants) | 3087 | 3035
  Change at Month 6 | 0.06 (0.777) | -0.33 (0.785)
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority; p < 0.0001, ANCOVA — P-value was based on analysis of covariance (ANCOVA) model with treatment and stratification variable (presence of established CV disease or CV risk factors without established CV disease) as factors, and baseline HbA1c, as a covariate; Least square (LS) Mean Difference (Net) = -0.39, 95% CI 2-sided [-0.43 to -0.35]

9. Secondary Outcome: Time From Randomization to Event of New Onset Renal Impairment or Worsening Existing Renal Impairment in All Participants
Description: New onset/worsening of existing renal impairment was first occurrence of any events: microalbuminuria and macroalbuminuria (albumin-to-creatinine ratio [ACR] >=30mcg/mg and ACR>=300 mcg/mg in spot urine), worsening albuminuria (microalbuminuria at Baseline developed macroalbuminuria, ACR increased >=30% from Baseline during treatment), newly developed chronic kidney disease (CKD) (eGFR >=90 milliliter per minute per 1.73 [mL/min/1.73]body surface area (BSA) and without kidney damage at Baseline changed to CKD Stage 1/higher as per National Kidney Foundation [NKF] Guidelines [2002]) or worsening of CKD (CKD Stage 1/higher as per NKF Guidelines [2002] worsened to higher CKD stages during treatment), or doubling of serum creatinine (creatinine value at least 2 times Baseline value and >=1.5 mg/dL during treatment.), or any of the following: end-stage renal disease, renal transplant, renal death. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The ITT set included all randomized participants regardless of whether they took study drug or not. This set was the same as the full analysis set.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 6000 | 6000
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.0054, Primary Analytic Method; Hazard Ratio (HR) = 0.869, 95% CI 2-sided [0.787 to 0.959]

10. Secondary Outcome: Time From Randomization to Event of New Onset Renal Impairment or Worsening Existing Renal Impairment in Participants With Prediabetes at Baseline
Description: New onset/worsening of existing renal impairment was first occurrence of any events: microalbuminuria and macroalbuminuria (ACR >=30mcg/mg and ACR >=300 mcg/mg in spot urine), worsening albuminuria (microalbuminuria at baseline developed macroalbuminuria, ACR increased >=30% from baseline during treatment), CKD (eGFR >=90 mL/min/1.73 BSA and without kidney damage at baseline changed to CKD Stage 1/higher as per NKF Guidelines [2002]) or worsening of CKD (CKD Stage 1/higher as per NKF Guidelines [2002] worsened to higher CKD stages during treatment), or doubling of serum creatinine (creatinine value at least 2 times baseline value and >=1.5 mg/dL during treatment.), or any of the following: end-stage renal disease, renal transplant, renal death. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 1976 | 2015
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio on a Cox regression model including treatment as covariate; p = 0.3661, Primary Analytic Method; Hazard Ratio (HR) = 0.904, 95% CI 2-sided [0.727 to 1.125]

11. Secondary Outcome: Time From Randomization to Event of New Onset Renal Impairment or Worsening Existing Renal Impairment in Participants With T2DM at Baseline
Description: New onset/worsening of existing renal impairment was first occurrence of any events: microalbuminuria and macroalbuminuria (ACR >=30 mcg/mg and ACR >=300 mcg/mg in spot urine), worsening albuminuria (microalbuminuria at baseline developed macroalbuminuria, ACR increased >=30% from baseline during treatment), CKD (eGFR >=90 mL/min/1.73 BSA and without kidney damage at baseline changed to CKD Stage 1/higher as per NKF Guidelines [2002]) or worsening of CKD (CKD Stage 1/higher as per NKF Guidelines [2002] worsened to higher CKD stages during treatment), or doubling of serum creatinine (creatinine value at least 2 times baseline value and >=1.5 mg/dL during treatment.), or any of the following: end-stage renal disease, renal transplant, renal death. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The T2DM analysis set included all participants in the ITT set who had T2DM at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 3403 | 3362
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority; p = 0.0082, Primary Analytic Method; Hazard Ratio (HR) = 0.855, 95% CI 2-sided [0.762 to 0.960]

12. Secondary Outcome: Time From Randomization to Event of Improvement in Renal Function in Participants With T2DM at Baseline
Description: Improvement in renal function was defined as first occurrence of regression of albuminuria or regression of CKD. Regression of albuminuria was defined as when participants with macroalbuminuria at baseline developed microalbuminuria or nonalbuminuria (ACR <30 mcg/mg in spot urine), or participants with microalbuminuria at baseline became nonalbuminuric, and ACR value decreased >= 30% from previous assessment during treatment. Regression of CKD defined as when participants with CKD Stage 1 or higher at baseline improved to normal or lower stages by NKF guidelines (eGFR >=90 with albuminuria at baseline improved to eGFR >=90 without albuminuria, or eGFR 60 to 89 at baseline became eGFR >=90 with or without albuminuria, or eGFR between 30 to 59 at baseline improved to >60 mL/min/1.73 BSA) during treatment. The outcome data was assessed using Kaplan-Meier estimate and Greenwood Formula.
Time Frame: Baseline up to end of study (Month 56)
Population: The T2DM analysis set included all participants in the ITT set who had T2DM at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 3403 | 3362
days | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants. | NA [NA to NA] — Median time and 95% confidence interval could not be calculated since quartile was not estimable due to higher number of censored participants.
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority — Hazard ratio was based on Cox-regression model including treatment and CV strata as covariates; p = 0.0297, Primary Analytic Method; Hazard Ratio (HR) = 1.182, 95% CI 2-sided [1.017 to 1.375]

13. Secondary Outcome: Percentage of Participants Who Met FDA-Defined Valvulopathy in Echocardiographically Determined Heart Valve Changes
Time Frame: Months 6 and 12
Population: The FDA-defined valvulopathy analysis set included all participants in the ITT set without FDA-defined valvulopathy at baseline. The FDA-defined valvulopathy analysis set where data was available at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 1935 | 1925
percentage of participants
  Month 6: number analyzed (Participants) | 1683 | 1681
  Month 6 | 1.4 | 2.1
  Month 12: number analyzed (Participants) | 1564 | 1579
  Month 12 | 1.5 | 1.8
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority; p = 0.5015, Regression, Logistic — P-value was based on logistic regression including treatment as a factor and baseline body mass index (BMI) as a covariate; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.69 to 2.11]

14. Secondary Outcome: Percentage of Participants With FDA-Defined Valvulopathy at Baseline Who Demonstrated Worsened FDA-Defined Valvulopathy
Time Frame: Months 6 and 12
Population: The ITT analysis set in participants with FDA-defined valvulopathy at baseline was used. The ITT analysis set in participants with FDA-defined valvulopathy at baseline where data was available at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 228 | 225
percentage of participants
  Month 6: number analyzed (Participants) | 194 | 201
  Month 6 | 2.1 | 3.5
  Month 12: number analyzed (Participants) | 180 | 189
  Month 12 | 1.7 | 2.1
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority; p = 0.7249, Regression, Logistic — P-value was based on logistic regression including treatment as a factor and baseline BMI as a covariate; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.29 to 5.98]

15. Secondary Outcome: Change From Baseline in Echocardiographically-Determined Pulmonary Arterial Systolic Pressure
Time Frame: Baseline, Month 12
Population: The ITT analysis set-participants in ECHO substudy included all randomized participants regardless of whether they took study drug or not. The ITT analysis set-participants in the ECHO substudy, where data was available at specified time points.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Lorcaserin 10 mg
Number analyzed (Participants) | 2167 | 2151
Millimeter of mercury (mmHg)
  Baseline: number analyzed (Participants) | 1368 | 1358
  Baseline | 26.4354 (7.66312) | 26.2029 (7.54123)
  Change at Month 12: number analyzed (Participants) | 882 | 893
  Change at Month 12 | -0.6418 (6.81716) | -0.8223 (7.23770)
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin 10 mg; Test type: Superiority; p = 0.2976, Mixed-effects model — P value was based on a mixed-effects model (unstructured covariance matrix) with repeated measures with treatment, month and treatment by month interaction as factors and baseline pulmonary arterial systolic pressure and baseline BMI as covariates; Least square (LS) Mean Difference (Net) = -0.9036, 95% CI 2-sided [-1.2908 to -0.5163]

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days after last dose of study drug (approximately 56 months)
Description: Adverse events were collected for the participants who were in the safety analysis set (all participants who received at least 1 dose of study drug and had at least one post dose safety assessment).
Arm/Group | Placebo | Lorcaserin 10 mg
All-Cause Mortality (participants affected / at risk) | 202/5992 | 219/5995
Serious Adverse Events (participants affected / at risk) | 2021/5992 | 1974/5995
Other Adverse Events (participants affected / at risk) | 4788/5992 | 4946/5995
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5992) | Lorcaserin 10 mg (N=5995)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 19 (19) | 12 (14)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 14 (14) | 11 (11)
Acute left ventricular failure (Cardiac disorders) | 3 (3) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 117 (131) | 105 (118)
Angina pectoris (Cardiac disorders) | 123 (136) | 142 (152)
Angina unstable (Cardiac disorders) | 106 (115) | 113 (129)
Anginal equivalent (Cardiac disorders) | 2 (2) | 2 (2)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 4 (4) | 6 (6)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 9 (9)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 102 (122) | 105 (120)
Atrial flutter (Cardiac disorders) | 22 (28) | 21 (23)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Atrioventricular block (Cardiac disorders) | 0 (0) | 4 (4)
Atrioventricular block complete (Cardiac disorders) | 7 (7) | 4 (4)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 7 (7)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 17 (17) | 18 (18)
Bundle branch block bilateral (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 2 (2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 19 (19) | 17 (17)
Cardiac discomfort (Cardiac disorders) | 7 (7) | 3 (3)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 21 (25) | 18 (19)
Cardiac failure acute (Cardiac disorders) | 5 (6) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 106 (139) | 91 (124)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 6 (6) | 7 (7)
Cardiogenic shock (Cardiac disorders) | 5 (5) | 4 (4)
Cardiomyopathy (Cardiac disorders) | 4 (4) | 5 (5)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 2 (2) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 3 (3)
Cor pulmonale acute (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 78 (80) | 87 (92)
Coronary artery occlusion (Cardiac disorders) | 6 (6) | 8 (10)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 13 (13) | 17 (17)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Hyperdynamic left ventricle (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 4 (4) | 3 (3)
Kounis syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Left atrial dilatation (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 3 (3)
Left ventricular failure (Cardiac disorders) | 2 (3) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 1 (13)
Mitral valve disease (Cardiac disorders) | 2 (2) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 12 (12) | 12 (12)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 31 (31) | 36 (38)
Myocardial ischaemia (Cardiac disorders) | 16 (17) | 14 (14)
Palpitations (Cardiac disorders) | 5 (5) | 6 (6)
Pericardial cyst (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 4 (6)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 2 (2)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 2 (3) | 3 (3)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 6 (6) | 15 (17)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 9 (9) | 11 (11)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 5 (5)
Tricuspid valve incompetence (Cardiac disorders) | 7 (7) | 6 (6)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 8 (8) | 3 (4)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 22 (27) | 13 (14)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 2 (3)
Choledochal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Microgenia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 8 (8) | 9 (9)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 5 (5)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 5 (5)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 2 (2)
Charles Bonnet syndrome (Eye disorders) | 0 (0) | 1 (1)
Deformity of orbit (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Oscillopsia (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular thrombosis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Vitreous adhesions (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal fat apron (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 10 (10) | 7 (7)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 6 (6)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (3) | 0 (0)
Coeliac artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 8 (8) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 8 (9)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 8 (8)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 4 (4) | 6 (6)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 4 (4)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterocele (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 5 (5) | 5 (5)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 6 (7) | 6 (6)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 27 (30) | 29 (29)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (10) | 11 (11)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 2 (2)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 9 (9) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 7 (7)
Intestinal perforation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (3) | 5 (5)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (9) | 2 (2)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 8 (8)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Omental infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 14 (15) | 13 (14)
Pancreatitis acute (Gastrointestinal disorders) | 15 (17) | 9 (9)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (6) | 8 (8)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 18 (22) | 11 (16)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 7 (7) | 6 (6)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 3 (3)
Uvulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Visceroptosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (7)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 5 (5) | 9 (10)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 7 (7) | 6 (6)
Chest pain (General disorders) | 21 (22) | 16 (16)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (2)
Death (General disorders) | 12 (12) | 16 (16)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 2 (2) | 3 (3)
Gastrointestinal complication associated with device (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Hernia pain (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Implant site erosion (General disorders) | 0 (0) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 132 (153) | 133 (164)
Oedema peripheral (General disorders) | 4 (4) | 4 (4)
Pain (General disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 2 (2)
Sudden death (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 2 (2)
Vascular stent occlusion (General disorders) | 1 (1) | 1 (1)
Vascular stent restenosis (General disorders) | 2 (2) | 3 (5)
Vascular stent thrombosis (General disorders) | 0 (0) | 2 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 2 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 14 (14) | 10 (10)
Cholecystitis acute (Hepatobiliary disorders) | 14 (14) | 12 (12)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 24 (25) | 14 (14)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 4 (4)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic vascular thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 4 (4) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 3 (3) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 2 (2) | 3 (3)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Abscess of salivary gland (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 9 (9) | 9 (9)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 2 (2)
Arthritis infective (Infections and infestations) | 2 (3) | 1 (1)
Bacteraemia (Infections and infestations) | 6 (6) | 3 (3)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 2 (2) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 26 (26) | 18 (19)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 71 (81) | 48 (52)
Cellulitis pasteurella (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 1 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 2 (3)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 4 (4)
Colonic abscess (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 7 (8) | 4 (4)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 1 (1)
Diabetic gangrene (Infections and infestations) | 2 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 17 (22) | 23 (26)
Emphysematous cystitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 4 (4)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 2 (2) | 1 (1)
Escherichia sepsis (Infections and infestations) | 2 (2) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Extradural abscess (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 13 (13) | 10 (10)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 7 (7)
Groin abscess (Infections and infestations) | 1 (1) | 1 (1)
Groin infection (Infections and infestations) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Human anaplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Human ehrlichiosis (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 3 (4) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (3) | 3 (4)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 10 (10) | 12 (12)
Kidney infection (Infections and infestations) | 2 (2) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 5 (6) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 2 (2) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 13 (14) | 11 (12)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 86 (90) | 92 (105)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 4 (4) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 2 (2) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 5 (5)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 4 (4) | 6 (6)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 1 (1)
Respiratory moniliasis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0)
Rocky mountain spotted fever (Infections and infestations) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 27 (27) | 37 (39)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Septic arthritis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Septic embolus (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 5 (5) | 7 (7)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal infection (Infections and infestations) | 3 (3) | 6 (6)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 40 (41) | 30 (30)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 7 (7) | 13 (13)
Vascular stent infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
West Nile viral infection (Infections and infestations) | 0 (0) | 2 (2)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 4 (4) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 4 (5)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 15 (17) | 21 (21)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 10 (11)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Humerus fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Joint capsule rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Kidney contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Pelvic fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 6 (7)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 9 (9) | 9 (9)
Road traffic accident (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 7 (8) | 5 (5)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 1 (1)
Aortic bruit (Investigations) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 1 (1)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
ECG signs of myocardial ischaemia (Investigations) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Heart rate decreased (Investigations) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio abnormal (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 3 (3)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Pulmonary arterial pressure increased (Investigations) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 8 (8) | 6 (6)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cholesterosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 21 (21) | 13 (14)
Diabetes mellitus (Metabolism and nutrition disorders) | 13 (13) | 11 (11)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 (5) | 5 (7)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Gout (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (11) | 6 (6)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 18 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6) | 10 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 12 (12) | 12 (12)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 11 (11) | 7 (7)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (26) | 25 (26)
Arthritis (Musculoskeletal and connective tissue disorders) | 16 (19) | 19 (20)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 16 (16)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 15 (15) | 6 (6)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 13 (13) | 12 (12)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 109 (121) | 93 (97)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 10 (11) | 5 (5)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 10 (10)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 11 (11)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Choroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 9 (9)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 4 (4)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 13 (13)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (21) | 20 (24)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 5 (5)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant sweat gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Mucinous cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 51 (51) | 50 (50)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (6)
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1)
Bickerstaff's encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 3 (3) | 2 (2)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 2 (2)
Brain stem stroke (Nervous system disorders) | 3 (3) | 0 (0)
Carotid artery disease (Nervous system disorders) | 2 (2) | 3 (3)
Carotid artery occlusion (Nervous system disorders) | 2 (2) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 17 (19) | 15 (15)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 4 (4) | 9 (9)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 41 (42) | 29 (31)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 2 (2)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve palsies multiple (Nervous system disorders) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 2 (2) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 9 (9) | 14 (14)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 2 (2)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 2 (2) | 3 (3)
Encephalopathy (Nervous system disorders) | 2 (2) | 4 (4)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 2 (2)
Frontal lobe epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 9 (10) | 5 (5)
Hemiparesis (Nervous system disorders) | 2 (2) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Hypertensive encephalopathy (Nervous system disorders) | 2 (2) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 3 (3)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 14 (14) | 13 (14)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 3 (3) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 4 (4) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (2)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 5 (6)
Migraine (Nervous system disorders) | 5 (5) | 5 (5)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 1 (1)
Myelomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 3 (3)
Nerve root compression (Nervous system disorders) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Parkinson's disease (Nervous system disorders) | 2 (2) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 13 (13) | 9 (9)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 7 (7) | 2 (2)
Seizure (Nervous system disorders) | 4 (4) | 10 (13)
Serotonin syndrome (Nervous system disorders) | 3 (4) | 3 (3)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Slow speech (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord disorder (Nervous system disorders) | 0 (0) | 2 (2)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 9 (9)
Superficial siderosis of central nervous system (Nervous system disorders) | 1 (1) | 0 (0)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 49 (51) | 54 (62)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 2 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 38 (39) | 46 (55)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 4 (4)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Vertebral artery dissection (Nervous system disorders) | 1 (1) | 1 (1)
Vertebral artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device failure (Product Issues) | 2 (2) | 0 (0)
Device loosening (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 2 (3)
Device pacing issue (Product Issues) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (2) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 12 (12)
Delirium (Psychiatric disorders) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 2 (2)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 6 (6) | 10 (12)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 1 (1)
Somatic delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 9 (9)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 57 (64) | 57 (61)
Acute prerenal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 3 (3) | 0 (0)
Bladder necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 7 (10) | 5 (6)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 18 (18) | 11 (11)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 2 (2)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal colic (Renal and urinary disorders) | 2 (2) | 5 (5)
Renal failure (Renal and urinary disorders) | 3 (3) | 4 (4)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterocele (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 6 (6) | 7 (7)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (9) | 6 (6)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 3 (4)
Adnexa uteri mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 10 (12) | 7 (11)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Mastoptosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Orchitis noninfective (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penis disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Priapism (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Scrotal haematocoele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 35 (37)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 12 (15)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 43 (53) | 39 (58)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 (40) | 27 (27)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 5 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (10)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 12 (13)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (6)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 20 (21)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 14 (14)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 14 (15)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Excessive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Convalescent (Social circumstances) | 1 (1) | 0 (0)
Spousal abuse (Social circumstances) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 2 (2) | 4 (4)
Aortic aneurysm (Vascular disorders) | 11 (11) | 6 (6)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 7 (7) | 14 (15)
Arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 13 (16) | 12 (12)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 14 (19) | 10 (10)
Hypertensive crisis (Vascular disorders) | 7 (7) | 8 (8)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 10 (10) | 16 (16)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Iliac artery disease (Vascular disorders) | 0 (0) | 1 (2)
Intermittent claudication (Vascular disorders) | 2 (2) | 6 (6)
Ischaemia (Vascular disorders) | 2 (2) | 0 (0)
Leriche syndrome (Vascular disorders) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1) | 2 (2)
Malignant hypertension (Vascular disorders) | 3 (3) | 1 (1)
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 5 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (11) | 14 (15)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 4 (4) | 2 (3)
Peripheral artery stenosis (Vascular disorders) | 4 (7) | 3 (4)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 7 (7) | 6 (6)
Peripheral venous disease (Vascular disorders) | 0 (0) | 2 (2)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0)
Reperfusion injury (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5992) | Lorcaserin 10 mg (N=5995)
Constipation (Gastrointestinal disorders) | 248 (268) | 336 (362)
Diarrhoea (Gastrointestinal disorders) | 324 (362) | 419 (478)
Nausea (Gastrointestinal disorders) | 286 (329) | 356 (398)
Fatigue (General disorders) | 302 (329) | 496 (548)
Oedema peripheral (General disorders) | 340 (385) | 267 (294)
Bronchitis (Infections and infestations) | 468 (584) | 455 (536)
Nasopharyngitis (Infections and infestations) | 338 (418) | 353 (426)
Upper respiratory tract infection (Infections and infestations) | 567 (690) | 528 (659)
Urinary tract infection (Infections and infestations) | 400 (575) | 440 (593)
Arthralgia (Musculoskeletal and connective tissue disorders) | 452 (542) | 457 (544)
Back pain (Musculoskeletal and connective tissue disorders) | 452 (496) | 457 (496)
Dizziness (Nervous system disorders) | 340 (407) | 537 (640)
Headache (Nervous system disorders) | 274 (316) | 383 (445)
Cough (Respiratory, thoracic and mediastinal disorders) | 303 (351) | 376 (431)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 310 (347) | 285 (312)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT02019264/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02019264/SAP_001.pdf